CLINICAL TRIAL: NCT03219580
Title: The Role of 5-Fluorouracil in Post-Operative Scar Formation Following Direct Brow Ptosis Repair
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eyelid and Facial Consultants (Other)
Collaborators: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LSUIRB#9586
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Brow Ptosis; Facial Scarring
MeSH Terms: interventions — Fluorouracil

STUDY DESIGN:
Intervention Model Description: Patients who undergo bilateral direct brow ptosis repair will be randomized to have one brow as the placebo arm and one arm as the active treatment arm. This original randomization will be maintained throughout the study.
Who Masked: Participant, Investigator
Masking Description: Both patients and physicians are blinded in this study. The study log is maintained by a study nurse who maintains the log of which side is randomized to placebo and active treatment arm respectively. The study nurse is also responsible for preparing the 2 arms in identical syringes, ensuring each arm is injected into its respective laterality
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5-Fluorouracil Active Treatment Arm (Active Comparator): A patient who has undergone bilateral direct brow ptosis repair and has elected to participate in the study will first have each of their brows randomized to either be the active treatment arm or the placebo arm. The active treatment arm brow will be injected with 0.05ml of 5-Fluorouracil 50mg/ml in several injections evenly spaced over the brow incision for a total of 0.3-0.6ml, repeated every three weeks for a total of 4 series of injections.
  Interventions: Drug: 5-Fluorouracil
- Placebo Arm (Placebo Comparator): A patient who has undergone bilateral direct brow ptosis repair and has elected to participate in the study will first have each of their brows randomized to either be the active treatment arm or the placebo arm. The placebo arm brow will be injected with 0.05ml of 0.9% Normal Saline in several injections evenly spaced over the brow incision for a total of 0.3-0.6ml, repeated every three weeks for a total of 4 series of injections.
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution

INTERVENTIONS:
Drug: 5-Fluorouracil — 50mg/ml concentration of 5-Fluorouracil to be injected intra-dermally in direct brow skin incisions
  Arms: 5-Fluorouracil Active Treatment Arm
Drug: Normal Saline Flush, 0.9% Injectable Solution — 0.9% concentration of Normal Saline Injectable Solution to be injected intra-dermally in direct brow skin incisions
  Arms: Placebo Arm

SUMMARY:
This is a double (physician and patient) blinded randomized controlled clinical trial in which patients who have undergone bilateral direct brow ptosis repair undergo a trial in which one of brow is injected with placebo 0.9% Normal Saline and the contra-lateral brow is injected with 0.3-0.6 mL over the entire brow of 50mg/mL 5-Fluorouracil sub-dermal injections. The researchers aim to investigate whether injecting 5-Fluorouracil preemptively will not only accelerate wound healing and decrease hypertrophic scar formation compared to placebo, but also improve overall scar appearance in a safe manner.

DETAILED DESCRIPTION:
In this double-blinded (physician and patient) randomized controlled clinical trial, the patient's left and right brows are randomized to either the placebo or treatment arm of the study and maintain this designation for the entirety of the study. This randomization is performed and recorded by the study nurse in the physician's office. This study nurse also will be responsible for preparing the placebo 0.9% Normal Saline (0.9%NS) and the 50mg/mL 5-Fluorouracil (5-FU). Both placebo and 5-FU are placed into identical syringes with 30 gauge needles, both materials are identical in color and clarity, making it impossible for physician or patient to correctly identify which injection is which without a label. Only the study nurse will be aware of which injection is which, and the nurse will ensure that the correct injection is placed into the correct brow at each visit via the study log that the nurse maintains.

A patient who has undergone bilateral direct brow ptosis repair who has agreed to participate in the study will first return for the post-operative day 10 visit where sutures are removed from the brow incisions. The patient returns on post-operative week three for their first injections, the details of which are below:

Starting on post-operative week three, the patient will receive 0.05mL aliquots of each injection (0.9%NS and 5-FU) sub-dermally into the brow incision spread out evenly over the brow, totaling 0.3-0.6 mL of each injection over each respective brow. Photos of the patient's brows will be taken, and then both the physician and patient will fill out a survey recording their impressions, the contents of which are listed in subsequent sections of this protocol. This same procedure will be repeated every three weeks for a total of up to four rounds of injections, thus the final round of injections will be given on post-operative week twelve. At each of these post-operative visits, incidence of any side effects is recorded, and if an unacceptably high rate of side effects occurs, the study will be precociously terminated.

At post-operative week fifteen, the blind is broken, and again photos are taken and physician and patient impressions are recorded via survey. After the blind is broken, if desired, the patient can opt to undergo a similar series of injections on the placebo arm of 5-FU.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone bilateral direct brow ptosis repair (either cosmetic of functional)

Exclusion Criteria:

* Known prior knowledge of the study's existence
* History of hypertrophic scarring
* Prior brow surgery, prior incisions or trauma to the forehead, brow or peri-ocular area in the past
* Patients who are decisionally or mentally impaired as they will be required to fill out the supplied survey and have the capacity for consent for the treatment
* Patients with any disease which may affect the brow (e.g. Myasthenia Gravis)
* Actively being treated for malignancy
* Uncontrolled autoimmune diseases with skin involvement

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall appearance | 1 year
  Patient and physician impression of overall appearance of the direct brow incision scar
Skin tone match | 1 year
  Patient and physician impression of how close the direct brow incision scar matches the patient's natural skin tone/color
Scar roughness/tough to touch | 1 year
  Patient and physician impression as to the degree of rough to the touch (ie fibrosis) is present in the direct brow incision scar
Scar is flush with eyebrow | 1 year
  Patient and physician impressions as to degree that direct brow incision scar is flush with skin of the brow

SECONDARY OUTCOMES:
Incidence of side effects | 1 year
  Any incidence of any side effects

CONTACTS AND LOCATIONS:
Overall Officials: Adham B. al Hariri, M.D., Principal Investigator — Eyelid and Facial Consultants New Orleans
Locations (2):
- United States (2):
  - Leonard J. Chabert Medical Center, Houma, Louisiana
  - Eyelid and Facial Consultants, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wendling J, Marchand A, Mauviel A, Verrecchia F. 5-fluorouracil blocks transforming growth factor-beta-induced alpha 2 type I collagen gene (COL1A2) expression in human fibroblasts via c-Jun NH2-terminal kinase/activator protein-1 activation. Mol Pharmacol. 2003 Sep;64(3):707-13. doi: 10.1124/mol.64.3.707. PMID 12920208
- [Background] Yoo DB, Azizzadeh B, Massry GG. Injectable 5-FU with or without added steroid in periorbital skin grafting: initial observations. Ophthalmic Plast Reconstr Surg. 2015 Mar-Apr;31(2):122-6. doi: 10.1097/IOP.0000000000000214. PMID 25025385
- [Background] Poetschke J, Gauglitz GG. Current options for the treatment of pathological scarring. J Dtsch Dermatol Ges. 2016 May;14(5):467-77. doi: 10.1111/ddg.13027. PMID 27119465
- [Background] Gupta S, Kalra A. Efficacy and safety of intralesional 5-fluorouracil in the treatment of keloids. Dermatology. 2002;204(2):130-2. doi: 10.1159/000051830. PMID 11937738
- [Background] Kontochristopoulos G, Stefanaki C, Panagiotopoulos A, Stefanaki K, Argyrakos T, Petridis A, Katsambas A. Intralesional 5-fluorouracil in the treatment of keloids: an open clinical and histopathologic study. J Am Acad Dermatol. 2005 Mar;52(3 Pt 1):474-9. doi: 10.1016/j.jaad.2004.09.018. PMID 15761426
- [Background] Fang QQ, Chen CY, Zhang MX, Huang CL, Wang XW, Xu JH, Wu LH, Zhang LY, Tan WQ. The Effectiveness of Topical Anti-scarring Agents and a Novel Combined Process on Cutaneous Scar Management. Curr Pharm Des. 2017;23(15):2268-2275. doi: 10.2174/1381612822666161025144434. PMID 27784253
- [Background] Khan MA, Bashir MM, Khan FA. Intralesional triamcinolone alone and in combination with 5-fluorouracil for the treatment of keloid and hypertrophic scars. J Pak Med Assoc. 2014 Sep;64(9):1003-7. PMID 25823177
- [Background] Darougheh A, Asilian A, Shariati F. Intralesional triamcinolone alone or in combination with 5-fluorouracil for the treatment of keloid and hypertrophic scars. Clin Exp Dermatol. 2009 Mar;34(2):219-23. doi: 10.1111/j.1365-2230.2007.02631.x. Epub 2008 Nov 6. PMID 19018794
- [Background] Huang L, Cai YJ, Lung I, Leung BC, Burd A. A study of the combination of triamcinolone and 5-fluorouracil in modulating keloid fibroblasts in vitro. J Plast Reconstr Aesthet Surg. 2013 Sep;66(9):e251-9. doi: 10.1016/j.bjps.2013.06.004. Epub 2013 Jun 28. PMID 23810214
- [Background] Pomerantz H, Hogan D, Eilers D, Swetter SM, Chen SC, Jacob SE, Warshaw EM, Stricklin G, Dellavalle RP, Sidhu-Malik N, Konnikov N, Werth VP, Keri J, Lew R, Weinstock MA; Veterans Affairs Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial Group. Long-term Efficacy of Topical Fluorouracil Cream, 5%, for Treating Actinic Keratosis: A Randomized Clinical Trial. JAMA Dermatol. 2015 Sep;151(9):952-60. doi: 10.1001/jamadermatol.2015.0502. PMID 25950503
- [Background] Jones CD, Guiot L, Samy M, Gorman M, Tehrani H. The Use of Chemotherapeutics for the Treatment of Keloid Scars. Dermatol Reports. 2015 May 21;7(2):5880. doi: 10.4081/dr.2015.5880. eCollection 2015 May 21. PMID 26236447